CLINICAL TRIAL: NCT02523924
Title: Pilot Study of 18F-DCFPyL PET/CT in the Evaluation of Men With an Elevated PSA Following Radical Prostatectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: J1545; IRB00062296 (Other: JHMIRB)
Record Dates: First submitted 2015-05-28; First posted 2015-08-14 (Estimated); Results first posted 2020-01-31 (Actual); Last update posted 2020-01-31 (Actual); Status verified 2020-01

CONDITIONS: Adenocarcinoma of the Prostate
MeSH Terms: interventions — 2-(3-(1-carboxy-5-((6-fluoropyridine-3-carbonyl)amino)pentyl)ureido)pentanedioic acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 18F-DCFPyL PET/CT (Experimental): Men with an elevated PSA following radical prostatectomy imaged with 18F-DCFPyL PET/CT
  Interventions: Drug: 18F-DCFPyL

INTERVENTIONS:
Drug: 18F-DCFPyL — 18F-DCFPyL PET/CT

SUMMARY:
This pilot study aims to investigate the diagnostic utility of 18F-DCFPyL, a novel low-molecular weight PSMA PET/CT imaging agent, in men with an elevated PSA following radical prostatectomy.

DETAILED DESCRIPTION:
18F-DCFPyL is a novel low-molecular weight PSMA imaging agent. A recent study of patients with metastatic prostate cancer found that PSMA PET/CT identified more sites of disease than conventional imaging with CT, MRI and bone scan. In this study we aim to investigate 18F-DCFPyL PET/CT in patients with an elevated PSA following radical prostatectomy. During the course of this study, patients will undergo two 18F-DCPyL PET/CT scans. The first scan will take place within 45 days of staging imaging and the second will take place following six months of standard of care therapy.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* History of adenocarcinoma of the prostate treated with radical prostatectomy
* Serum PSA level ≥0.2 ng/mL at least 45 days prior to study enrollment
* Completed staging evaluation with bone scan as well as CT or MRI of the abdomen and pelvis at least 45 days prior to study enrollment

Exclusion Criteria:

* Intention to enroll in a blinded therapeutic clinical trial
* History of other malignancy diagnosed within the last three years (the exception of squamous cell or basal cell carcinoma of the skin)

Ages: 18 Years to 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2015-06-02 (Actual); Primary Completion 2016-11-04 (Actual); Study Completion 2019-03-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- SKCCC, Baltimore, Maryland, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 19 patients did not meet inclusion criteria.
Period: Overall Study
Arm/Group | 18F-DCFPyL PET/CT
Started | 31
Completed | 31
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | 18F-DCFPyL PET/CT
Number analyzed (Participants) | 31
Age, Continuous [Median (Full Range); unit: years] | 63 [45 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 31
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 27
  More than one race | 0
  Unknown or Not Reported | 4
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 31
Months since radical prostatectomy [Median (Full Range); unit: months] | 30 [4 to 152]
Gleason grade group [Count of Participants; unit: Participants] — The Gleason score ranges from 2-10 with a higher score reflecting less-differentiated tumors with worse prognosis. The total score is a sum of two numbers which are based on the microscopic appearance of cells. The first number is the score based on the dominant, cell morphology (scored 1-5) and the second number is based on the highest grade of the non-dominant cell pattern (scored 1-5)
  Participants
    1 | 2
    2 | 6
    3 | 13
    4 | 1
    5 | 9
Pathologic stage [Count of Participants; unit: Participants]
  pT2 | 11
  pT3a | 14
  pT3b | 6
Positive surgical margin [Count of Participants; unit: Participants] | 13
Prostate Specific Antigen (PSA) [Median (Full Range); unit: ng/mL] | 0.4 [0.2 to 28.3]

OUTCOME MEASURES:

1. Primary Outcome: Number of Putative Sites of Metastatic Disease as Determined by 18F-DCFPyL PET/CT
Description: Number of sites with 18F-DCFPyL uptake consistent with prostate cancer.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | 18F-DCFPyL PET/CT
Number analyzed (Participants) | 31
Participants
  at least 1 site | 21
  > 1 site | 5
  no sites | 5

2. Primary Outcome: Location of Putative Sites of Metastatic Disease as Determined by 18F-DCFPyL PET/CT
Description: Location of uptake of 18F-DCFPyL consistent with prostate cancer.
Time Frame: 6 months
Population: Location of 18F-DCFPyL uptake could only be assessed in patients with at least 1 site of 18F-DCFPyL uptake (26/31)
Measure: Count of Participants; unit: Participants
Arm/Group | 18F-DCFPyL PET/CT
Number analyzed (Participants) | 26
Participants
  Prostate bed | 8
  Pelvic lymph node | 14
  Nonpelvic lymph node | 2
  Bone | 2
  Viscera | 0

3. Secondary Outcome: Correlation of 18F-DCFPyL PET/CT Findings With Prostate Specific Antigen (PSA) Levels
Description: Number of participants with PSA 0.2-1.0ng/mL OR PSA >1.0ng/mL with at least 1 site of uptake of 18F-DCFPyL consistent with prostate cancer.
Time Frame: 6 months
Population: Only 22/31 participants had a PSA of 0.2-1.0ng/mL and 9/31 participants had PSA >1.0ng/mL.
Measure: Count of Participants; unit: Participants
Arm/Group | 18F-DCFPyL PET/CT
Number analyzed (Participants) | 31
Participants
  PSA 0.2-1.0 ng/mL: number analyzed (Participants) | 22
  PSA 0.2-1.0 ng/mL | 13
  PSA >1.0 ng/mL: number analyzed (Participants) | 9
  PSA >1.0 ng/mL | 8

4. Secondary Outcome: Correlation of Findings on 18FDCFPyL PET/CT With Those Found on Conventional Imaging (Bone Scan and Cross-sectional Imaging)
Description: Number of sites with uptake on 18F-DCFPyL PET/CT and corresponding lesions identified on conventional imaging.
Time Frame: 6 months
Population: Data was not collected for this outcome as participants did not have conventional imaging correlates.
Arm/Group | 18F-DCFPyL PET/CT
Number analyzed (Participants) | 0

5. Secondary Outcome: Correlation of Findings on 18F-DCFPyL PET/CT With Tissue Histology and PSMA Expression of Biopsied/Resected Pathology Specimens
Description: Number of sites with 18F-DCFPyL uptake from which biopsy specimens show PSMA expression.
Time Frame: 6 months
Population: Data was not collected to assess this outcome measure as confirmatory biopsy was not practical to perform and histopathologic confirmation is not available.
Arm/Group | 18F-DCFPyL PET/CT
Number analyzed (Participants) | 0

6. Other Pre Specified Outcome: Correlation of 18F-DCFPyL PET/CT Findings With Time to Disease Progression
Time Frame: 6 months
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Assessment of Treatment Response by 18F-DCFPyL PET/CT
Time Frame: 6 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | 18F-DCFPyL PET/CT
All-Cause Mortality (participants affected / at risk) | 0/31
Serious Adverse Events (participants affected / at risk) | 0/31
Other Adverse Events (participants affected / at risk) | 0/31

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-02-21): https://cdn.clinicaltrials.gov/large-docs/24/NCT02523924/Prot_SAP_000.pdf